CLINICAL TRIAL: NCT00941291
Title: Long-term Outcome of Idiopathic Macular Hole Surgery
Brief Title: Outcome of Idiopathic Macular Hole
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Professor Creuzot-Garcher Catherine
Other Study IDs: Macular hole 1
Record Dates: First submitted 2009-03-30; First posted 2009-07-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Idiopathic Macular Hole
Keywords: idiopathic macular hole; cataract; edema; Reopening
MeSH Terms: conditions — Cataract; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- vitrectomy in pseudophakic eyes
- vitrectomy and cataract:combined procedure
- vitrectomy followed by cataract extraction
- vitrectomy on phakic eyes

SUMMARY:
The purpose of this study is to evaluate the role of cataract surgery and cystoid macular edema (CME) on reopening of idiopathic macular holes (IMH).

ELIGIBILITY:
Inclusion Criteria:

* Patients with with stage 2, 3, or 4 Idiopathic Macular Hole after successful Idiopathic Macular Hole repair

Exclusion Criteria:

* All patients without stage 2, 3, or 4 Idiopathic Macular Hole repair

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and thirty patients (135 eyes) with stage 2, 3, or 4 IMH were included after successful IMH repair
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2002-01; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Long-term outcome of idiopathic macular hole surgery | 37 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Creuzot-Gracher, MD, PhD, Principal Investigator — Ophthalmology unit CHU Dijon
Locations (1):
- Ophthalmology Unit CHU Dijon, Dijon, Burgundy, France

REFERENCES:
- [Derived] Passemard M, Yakoubi Y, Muselier A, Hubert I, Guillaubey A, Bron AM, Berrod JP, Creuzot-Garcher C. Long-term outcome of idiopathic macular hole surgery. Am J Ophthalmol. 2010 Jan;149(1):120-6. doi: 10.1016/j.ajo.2009.08.003. Epub 2009 Oct 20. PMID 19846059